CLINICAL TRIAL: NCT00910884
Title: Stage IV Breast Cancer Gene Expression Control Using Micro-Trace and Plant Extracted Natural G.R.A.S. (Generally Accepted As Safe), Compounds in Adjunct Therapy Alongside Conventional Cancer Protocols
Brief Title: Plant Extracted Natural Compounds Impact on Stage IV Breast Cancer Survival Time and Remission.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brabant Research (Industry)
Responsible Party: Principal Investigator, Dr. Richard Lasker, Director, Brabant Research
Other Study IDs: CDR0000643461; BRABANT-00005271
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage III breast cancer; stage IV breast cancer; hormonal cancers; skin cancers
MeSH Terms: conditions — Breast Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm I: Patients receive oral GRAS supplements daily for 12 months or as possible within the patient's parameters.
  Interventions: Other: laboratory biomarker analysis; Procedure: therapeutic dietary intervention
- Arm II: Patients do not receive supplements.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — No supplements are given
Procedure: therapeutic dietary intervention — Given orally daily for 12 months
  Groups: Arm I

SUMMARY:
RATIONALE: Plant extracted natural compounds, in an adjunct therapy position, slow the growth and reproduction of Stage IV Breast Cancer tumor cells. May help eradicate different types of cancers.

PURPOSE: The purpose of this randomized Phase I trial is to first IDENTIFY, through laboratory analysis and validating cellular biochemical pathways, and HELP CONTROL, using natural plant extracted compounds, G.R.A.S. (Generally Accepted As Safe), compounds, the reproduction, growth progress and metastasis of Stage IV Breast Cancer cells. The therapy position is adjunct to conventional therapies and in "one-off" trials have been excitingly effective for long-term survival. Novel use of bioactive GRAS compounds to augment and enhance conventional cancer therapies and as stand-alone parallel therapies.

DETAILED DESCRIPTION:
OBJECTIVES:

To utilize multiple naturally-occurring bioalkaloids, bioactive "compounds of interest" from multiple sources, to influence prostate, breast, and uterine cancer pathways in cancer patients and cancer patients in remission. Other cancer types may be applicable.

To utilize specific naturally-occurring bioalkaloids and bioactive "compounds of interest" to suppress cancer proliferation-stimulation/growth activities induced by normal cancer metabolism including environmental estrogen impact, estrogen-mimicking compounds, estrogen-influencing and testosterone-type compounds.

To utilize DNA interaction with proliferating cancer cells via intercalation, which has a binding impact activity that then impairs DNA polymerase furthering DNA strand breakage and complete apoptosis. In addition, these bioactive compounds through intercalation, prevent cancer-cell DNA strand breakage from re-connection and repair, (limitlessness) while depleting nuclear topoisomerase, the enzyme also targeted by a number of conventional chemotherapy routes. Finally; a number of the bioalkaloids binds to cancer telomeres capping them at specific number or reducing them to "one and done."

Natural GRAS compounds, in previous studies that background this research, reduced secondary bonding of TMPRSS2-ERG fusing affecting testosterone & estrogen hormone influence in cell proliferation. Variant mRNAs of, for example, the TMPRSS2-ERG fusing pathway were affected whereas normalized mRNAs in all other cells were not, a mechanism and chemistry not readily understood.

To utilize natural extracted plant compounds as a means to influence DIABLO (direct inhibitor of apoptosis binding protein with low isoelectric point) by downregulating over 350 genes which influence extracellular matrix (ECM) receptor interaction, and complement coagulation cascades were upregulated.

To utilize applications of, or ingestion of, specifically grown plant species/subspecies, extract the "compounds of action" or "compounds of activity" but maintaining an "entourage-affect by protecting "multi-compound complex arrangement chemistry" to maintain normal metabolic functionality of the compounds of interest..

BACKGROUND DATA:

Pharmaceutica has, since the turn of the 1800s to the 1900s, tried to find, extract and/or synthesize plant & biological compounds that have the highest activity in a given medical treatment regime. In many cases the object was to get to the heart of the active compound, discarding non-active compounds,and, in other cases for various reasons including stockholder satisfaction, to be able to patent the synthesis chemistry and prevent duplication by competitors.

The one point of this important to this work is that the natural multi-compounds were the "compounds of action" for centuries and in most cases, in the natural form they were utilized in pre-20th century medicine, while the action of control was usually much slower, the side affects were non-existent.

Recent research (sic) now places a more important role of the "multi-compound" and the "entourage-effect' they have as cancer cells are quick to evolve, like viruses, and where the pharmaceutica "single compound of action" approach works well when ALL the cancer cells are eliminated, does not work well when surviving cells evolve to create resistance...a common outcome to most advanced stage cancers.

The "entourage-effect" using the "multi-compound" natural extracted compounds appears to negate the evolution/resistance response of cancerous cells by having multiple "chemistries of action" involved the cancer-control process which then hides/disguises the metabolic pathway of control from the surviving cancer cells.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: Patients receive oral natural supplements comprising indole-3-carbinol, perillyl alcohol, glucuronic acid, and flavonoids daily for 12 months. Patients also consume whole foods comprising indole-3-carbinol and a diet that eliminates exogenous growth hormones.

Arm II: Patients do not receive natural supplements or consume whole foods or a special diet.

Levels of compounds of interest are measured by inductively-coupled plasma mass spectrometry, high performance liquid chromatography, gas chromatography, and matrix-assisted laser desorption/ionization time of flight mass spectrometry.

After completion of study therapy, patients are followed periodically for 6 months and monitored for a second 6 months period.

1. Krimsky S (December 2001). "An epistemological inquiry into the endocrine disruptor thesis". Ann. N. Y. Acad. Sci. 948 (1): 130-42. doi:10.1111/j.1749-6632.2001.tb03994.x. PMID 11795392.
2. Marinucci L, Bodo M, Balloni S, Locci P, Baroni T. "Sub-Toxic Nicotine Concentrations Affect Extracellular Matrix and Growth Factor Signaling Gene Expressions in Human Osteoblasts." J Cell Physiol. 2014 Apr 29. doi: 10.1002/jcp.24661. PMID: 24777817
3. Camargo IC, Leite GA, Pinto T, Ribeiro-Paes JT. "Histopathologycal findings in the ovaries and uterus of albino female rats promoted by co-administration of synthetic steroids and nicotine." Exp Toxicol Pathol. 2014 Jul;66(4):195-202. doi: 10.1016/j.etp.2014.01.005. Epub 2014 Feb 18. PMID: 24556002
4. Raval AP. "Nicotine addiction causes unique detrimental effects on women's brains." J Addict Dis. 2011 Apr;30(2):149-58. doi: 10.1080/10550887.2011.554782. Review. PMID: 21491296
5. Holloway AC, Salomon A, Soares MJ, Garnier V, Raha S, Sergent F, Nicholson CJ, Feige JJ, Benharouga M, Alfaidy N. "Characterization of the adverse effects of nicotine on placental development: in vivo and in vitro studies." Am J Physiol Endocrinol Metab. 2014 Feb 15;306(4):E443-56. doi: 10.1152/ajpendo.00478.2013. Epub 2013 Dec 24. PMID: 24368670
6. Bavarva JH, Tae H, Settlage RE, Garner HR. "Characterizing the Genetic Basis for Nicotine Induced Cancer Development: A Transcriptome Sequencing Study." PLoS One. 2013 Jun 18;8(6):e67252. Print 2013. PMID: 23825647
7. Hayes, Tyrone B.; Anderson, Lloyd L.; Beasley, Val R.; de Solla, Shane R.; Iguchi, Taisen; et al. (2011). "Demasculinization and feminization of male gonads by atrazine: Consistent effects across vertebrate classes". The Journal of Steroid Biochemistry and Molecular Biology 127 (1-2): 64-73. doi:10.1016/j.jsbmb.2011.03.015. PMID 21419222
8. Atrazine: Chemical Summary. Toxicity and Exposure Assessment for Children's Health (Report). U.S. Environmental Protection Agency. 4/24/2007
9. Mizota, K.; Ueda, H. (2006). "Endocrine Disrupting Chemical Atrazine Causes Degranulation through Gq/11 Protein-Coupled Neurosteroid Receptor in Mast Cells". Toxicological Sciences 90 (2): 362-8. doi:10.1093/toxsci/kfj087. PMID 16381660
10. Thomas, Christoforos; Strom A.; Lindberg K.; Gustafsson J. (22 June 2010). "Estrogen receptor beta decreases survival of p53-defective cancer cells after DNA damage by impairing G2/M checkpoint signaling". Breast Cancer Research and Treatment 127 (2): 417-427. doi:10.1007/s10549-010-1011-z. PMID 20623183

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate, breast, or uterine cancer

  * Early or late stage disease
* Currently waiting to initiate conventional therapy or radiotherapy OR receiving concurrent conventional chemotherapy or radiation therapy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior or concurrent chemotherapy or hormonal therapy for cancer allowed

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female in breast cancer, any Stage.
Study Population: Breast cancer not limited to "in-remission only." Any Stage of cancer; preference in population to Stage IV.
  Inclusions:
  Breast Cancer, any stage. In remission or not. Uterine Cancer, any stage. In remission or not. Ovarian Cancer, any stage. In remission or not. Hormonal Cancers, cell division driven by hormones. In remission or not. Skin Cancers, any stage. In remission or not.
  Exclusions:
  None noted at this time. Exclusions may be modified upon presentation. Look for updates.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Utilize GRAS plant extracted compounds for suppression of cancer-cell replication. | 12 months
  Using adjunct therapy to augment and increase efficacy of conventional cancer treatments
Suppression of cancer genetic pathways to reproduction. | 6 months
  suppress cancer cell proliferation
Reduction of secondary bonding of TMPRSS2-ERG fusing using, among other modes of action, DPPH radical-scavenging activity | 6 months
  Monitor levels
Monitor normal metabolic function while measuring cancer-marker levels. | 6 months
  metabolic function testing

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Lasker, PhD, Principal Investigator — Brabant Research
Locations (1):
- Brabant Research, Incorporated, Spokane Valley, Washington, United States